CLINICAL TRIAL: NCT02262689
Title: A Randomised Placebo-controlled Study to Evaluate the Effects of GSK2256294 Following Repeat Dosing on Pulmonary Artery Pressure in Healthy Volunteers Under Normoxic and Hypoxic Conditions
Brief Title: To Evaluate Effects of GSK2256294 on Pulmonary Artery Pressure in Healthy Volunteers Under Normoxic and Hypoxic Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201402
Record Dates: First submitted 2014-10-09; First posted 2014-10-13 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: GSK2256294; normoxic; hypoxic; Pulmonary artery systolic pressure (PASP)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypoxia | interventions — N-((4-cyano-2-(trifluoromethyl)phenyl)methyl)-3-((4-methyl-6-(methylamino)-1,3,5-triazin-2-yl)amino)cyclohexanecarboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK2256294 15 mg (Experimental): Randomised subjects will be instructed to take three capsules of GSK2256294 15 mg, each morning for 7 days. Subjects will undergo echocardiography under normoxic and hypoxic conditions on Day 1 pre-dose and on Day 7 post-dose.
  Interventions: Drug: GSK2256294
- Placebo (Placebo Comparator): Randomised subjects will be instructed to take three capsules of matching placebo, each morning for 7 days. Subjects will undergo echocardiography under normoxic and hypoxic conditions on Day 1 pre-dose and on Day 7 post-dose.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK2256294 — GSK2256294 will be supplied as gelatin capsule to be administered orally with the unit dose 5 mg / dose level 15 mg
  Arms: GSK2256294 15 mg
Drug: Placebo — Matched Placebo will be supplied as gelatin capsule to be administered orally
  Arms: Placebo

SUMMARY:
The study evaluates the effect of GSK2256294 exposure at steady state on pulmonary artery systolic pressure (PASP) in healthy volunteers, under hypoxic conditions, after 7 days of dosing. It is single centre, double blind, randomized, placebo-controlled study to be conducted in approximately 30 healthy volunteers. Subjects will be screened no more than 30 days. Subject will be admitted in clinical unit on Day -1. Subject will be dosed for 7 days in unit in morning on all days except for dosing on Days 3 -6. Dosing on Days 3 -6 will occur at home. Subjects will return to the unit on the evening of Day 6 and remain there until Day 8. Subjects will undergo echocardiography under normoxic and hypoxic on Day 1 pre-dose and on Day 7 post-dose. Subject will be followed up for 28- 32 days after discharge. The maximum estimated time that a subject will be enrolled in the study is 62 days from the screening visit to follow up.

ELIGIBILITY:
Inclusion Criteria:

* AGE: Between 18 and 65 years of age inclusive, at the time of signing the informed consent
* Screening echocardiogram of at least good quality, without clinically significant abnormalities, and with mild-moderate tricuspid regurgitation sufficient for the reliable estimation of PASP, as determined by the echocardiography core laboratory or responsible cardiologist.
* Screening PASP within the normal range according to site standards
* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator [in consultation with the Medical Monitor if required] agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >= 60 kilogram and body mass index within the range 19 - 35 kilogram per square meter (inclusive)
* Female subject is eligible to participate if she is of non-reproductive potential defined as: Pre-menopausal females with one of the following: documented tubal ligation, documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion, hysterectomy, and documented bilateral oophorectomy. Postmenopausal criteria is defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause (refer to laboratory reference ranges for confirmatory levels)]; females on hormone replacement therapy (HRT) must discontinue their HRT before the start of the study; for those whose menopausal status is in doubt, they will be required to use one of the highly effective contraception methods and may need to have a blood sample taken to check FSH/estradiol levels.
* Male subjects with female partners of child bearing potential must comply with the following contraception requirements from the time of first dose of study medication until two weeks after the last dose of study medication; vasectomy with documentation of azoospermia; male condom plus partner use of one of the contraceptive options below: Contraceptive subdermal implant that meets the Standard Operating Procedure (SOP)effectiveness criteria including a <1% rate of failure per year, as stated in the product label, Intrauterine device or intrauterine system that meets SOP effectiveness criteria including a <1% rate of failure per year, as stated in the product label, Oral Contraceptive, either combined or progestogen alone, Injectable progestogen, Contraceptive vaginal ring; percutaneous contraceptive patches. These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.
* Capable of giving signed informed consent as described in protocol, which includes compliance with the requirements and restrictions listed in the consent form and in protocol

Exclusion Criteria:

* Subjects with sickle cell trait.
* History of pulmonary hypertension.
* Alanine aminotransferase (ALT) and bilirubin >1.5x Upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* QTcF > 450 milliseconds (msec) NOTE: The QTc is the QT interval corrected for heart rate according to Fridericia's formula (QTcF). The specific formula that will be used to determine eligibility and discontinuation for an individual subject should be determined prior to initiation of the study. In other words, several different formulae cannot be used to calculate the QTc for an individual subject and then the lowest QTc value used to include or discontinue the subject from the trial. For purposes of data analysis, QTcF will be used as specified in the Reporting and Analysis Plan (RAP).
* Permitted Medications and Non-Drug Therapies: Acetaminophen, at doses of =< 2 grams/day is permitted for use any time during the study. Other concomitant medication may be considered on a case by case basis by the investigator in consultation with the GSK Medical Monitor. All concomitant medications taken during the study will be recorded in the case report form. The minimum requirement is that drug name, dose administered and the dates of administration be recorded.
* Prohibited Medications and Non-Drug Therapies: Subjects must abstain from taking prescription or non-prescription drugs (including vitamins and dietary or herbal supplements), within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication until completion of the follow-up visit, unless in the opinion of the Investigator and sponsor the medication will not interfere with the study. - History of regular alcohol consumption within 6 months of the study defined as: For US sites: an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 grams of alcohol: 12 ounces (360 milliliter [ml]) of beer, 5 ounces (150 ml) of wine or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment. For potent immunosuppressive agents, subjects with presence of hepatitis B core antibody (HBcAb) should also be excluded.
* A positive pre-study drug/alcohol screen.
* A positive test for Human Immunodeficiency Virus (HIV) antibody.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within 56 days.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-01-08 (Actual); Primary Completion 2015-04-24 (Actual); Study Completion 2015-04-24 (Actual)

PRIMARY OUTCOMES:
Change from baseline of PASP under hypoxic conditions | Day 1 and Day 7
  PASP is an indicator of cardiac hemodynamic status and is non-invasively estimated by echocardiography. Change from baseline in PASP under hypoxic conditions following 7 days of GSK2256294 15 milligrams (mg) once daily. Change from baseline was calculated as the Day 7 value minus the Day1 value.

SECONDARY OUTCOMES:
Change from baseline of PASP under normoxic conditions | Day 1 and Day 7
  The PASP is an indicator of cardiac hemodynamic status and is non-invasively estimated by echocardiography. Change from baseline in PASP under normoxic conditions following 7 days of GSK2256294 15 mg once daily. Change from baseline was calculated as the Day 7 value minus Day 1 value.
Number of subjects with Adverse events (AEs) | Up to Day 32
  An AE is any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Assessment of 12-lead electrocardiogram (ECG) | Up to Day 32
  Triplicate 12-lead ECGs will be obtained at each time point using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QT duration corrected for heart rate by Fridericia's formula (QTcF) intervals
Assessment of vital sign measurements | Up to Day 32
  Vital sign assessments includes temperature, blood pressure (systolic and diastolic) and pulse rate. measurements
Assessment of physical examination findings | Up to Day 32
  A complete physical examination will include, at a minimum, assessment of the Cardiovascular, Respiratory, Gastrointestinal and Neurological systems. Height and weight will also be measured and recorded. A brief physical examination will include, at a minimum assessments of the lungs, cardiovascular system, and abdomen (liver and spleen).
Assessment of clinical laboratory parameters | Up to Day 32
  Clinical laboratory parameters includes haematology, clinical chemistry and urinalysis

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 201402 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/201402?search=study&b'search_terms=201402'#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 201402 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 201402 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 201402 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 201402 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 201402 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 201402 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 201402 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register